CLINICAL TRIAL: NCT00922714
Title: Glutamine to Intensive Care Patients - a Prospective, Double-Blind, Placebo-Controlled Multicenter Study in the Scandinavian Countries
Brief Title: Scandinavian Intensive Care Unit (ICU) Glutamine Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment, stopped after 4 years
Sponsor: Scandinavian Critical Care Trials Group (Other)
Responsible Party: Jan Wernerman, Karolinska University Hospital Huddinge
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Scandinavian Glutamin Study
Record Dates: First submitted 2009-06-15; First posted 2009-06-17 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: ICU Patients
Keywords: Glutamine; ICU patients; Critically ill; Nutrition
MeSH Terms: conditions — Critical Illness | interventions — Glutamine; alanylglutamine; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glutamine (Experimental): Intravenous glutamine supplementation (0.285 g/kg body weight/24 h)
  Interventions: Drug: Glutamine
- Control (Placebo Comparator): saline
  Interventions: Drug: saline (placebo)

INTERVENTIONS:
Drug: Glutamine — Intravenous glutamine supplementation (0.285 g/kg body weight/24 h)
  Other Names: L-alanyl-L-glutamine, Dipeptiven
  Arms: Glutamine
Drug: saline (placebo) — NaCl 0.9 g/L
  Arms: Control

SUMMARY:
This is a prospective double-blinded placebo-controlled block randomized study in intensive care patients comparing intravenous glutamine supplementation to placebo. The hypothesis is an improvement of clinical outcome. The primary endpoint is a reduction in the Sequential Organ Failure Assessment (SOFA) score on day 7 of treatment.

DETAILED DESCRIPTION:
This is a prospective double-blinded placebo-controlled block randomised study in intensive care patients comparing intravenous glutamine supplementation (0.285 g/kg body weight/24 h) to placebo. Inclusion criteria are patients treated for more than 3 days. Primary endpoint is a reduction in SOFA-score on day 7 of treatments. Secondary endpoints are: ICU-mortality, 6-months mortality, length of ICU stay, organ failure free days as well as reduction in SOFA-score on day 10 of treatment. Nutrition will be standardised so that not less than 80% of the target which is basal energy expenditure according to Harris & Benedict is given daily. Enteral nutrition is preferred, but a combination of enteral and parenteral nutrition is recommended to achieve the nutritional target. For statistical comparison non-parametric rank order statistics will be used. To detect a 0.75-point difference in the reduction of SOFA-score on day 7 of treatment, a total of 1,000 patients will be needed.

ELIGIBILITY:
Inclusion Criteria:

* admission to the ICU
* decision to give the patient full nutrition
* APACHE II score > 10 at admission
* age 18-85 years

Exclusion Criteria:

* readmission to the ICU after a previous ICU-stay in which the patient has been included into the study
* subjects with any condition which in the opinion of the attending physician makes the subject unsuitable for inclusion
* no informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2003-10; Primary Completion 2007-05 (Actual); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
A reduction in SOFA-score | Day 7 of treatment

SECONDARY OUTCOMES:
Mortality | ICU stay and 6 months
Length of ICU stay | ICU stay
Organ failure free days | ICU stay
Reduction in SOFA-score | Day 10 of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jan Wernerman, MD, PhD, Principal Investigator — Dept Anesthesiology and Intensive Care Medicine, KArolinska University Hospital Huddinge, Stockholm, Sweden
Locations (1):
- Intensive Care Unit, Karolinska University Hospital Huddinge, Stockholm, Sweden